CLINICAL TRIAL: NCT00706563
Title: A Phase III Study for Evaluation of Immunogenicity and Reactogenicity of Fluarix™ / Influsplit SSW® 2008/2009 in People Aged 18 Years or Above
Brief Title: A Study for Evaluation of Immunogenicity and Reactogenicity of Fluarix™ / Influsplit SSW® 2008/2009 in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 111631
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Results first posted 2009-08-25 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-07

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — fluarix

ARMS (2):
- Fluarix Adult Group (Experimental): Subjects who are 18-40 years of age received one dose of Fluarix™.
  Interventions: Biological: Fluarix™
- Fluarix Elderly Group (Experimental): Subjects who are ≥ 60 years of age received one dose of Fluarix™.
  Interventions: Biological: Fluarix™

INTERVENTIONS:
Biological: Fluarix™ — Single intramuscular dose on Day 0
  Other Names: Influsplit

SUMMARY:
This study is designed to test the immunogenicity and reactogenicity of the Fluarix™/Influsplit SSW® influenza vaccine containing the influenza strains recommended for the 2008-2009 season.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female aged 18 years or above at the time of the vaccination.
* Written informed consent obtained from the subject.
* Healthy subjects or with well-controlled chronic diseases as established by medical history and clinical examination before entering into the study.
* If the subject is female, she must be of non-childbearing potential or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for 2 months after completion of the vaccination series

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the vaccination or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the vaccine dose.
* Administration of immunoglobulins and/or any blood products within the three months preceding the administration of the study vaccine or planned during the study.
* Administration of an influenza vaccine within 1 year preceding the study start.
* Administration of an influenza vaccine other than the study vaccine during the entire study
* Clinically or virologically confirmed influenza infection within 1 year preceding the study start
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Acute disease at the time of enrolment.
* Acute clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Not stabilized or clinically serious chronic underlying disease.
* Lactating female.
* History of chronic alcohol consumption and/or drug abuse.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Any condition which, in the opinion of the investigator, prevents the subject from participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-07-07 (Actual); Primary Completion 2008-07-30 (Actual); Study Completion 2008-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Germany (2):
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Freital, Saxony

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 111631 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111631 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111631 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111631 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111631 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111631 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111631 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fluarix Adult Group | Fluarix Elderly Group
Started | 61 | 59
Completed | 61 | 59
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluarix Adult Group | Fluarix Elderly Group | Total
Number analyzed (Participants) | 61 | 59 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (13.26) | 68.8 (5.25) | 53.7 (18.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 34 | 70
  Male | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Hemagglutination Inhibition (HI) Antibody Titer
Description: Titers given as geometric mean titer (GMT) were presented for all three vaccine influenza virus strains
Time Frame: At Day 0 and 21
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Fluarix Adult Group | Fluarix Elderly Group
Number analyzed (Participants) | 61 | 59
titer
  A/Brisbane (Day 0) | 13.6 [10.1 to 18.2] | 11.6 [9.1 to 14.9]
  A/Brisbane (Day 21) | 165.5 [119.2 to 229.7] | 68.2 [48.4 to 96.3]
  A/Uruguay (Day 0) | 7.6 [6.2 to 9.3] | 9.7 [7.3 to 12.9]
  A/Uruguay (Day 21) | 90.7 [60.2 to 136.5] | 120.6 [76.1 to 191.0]
  B/Brisbane (Day 0) | 102.1 [74.4 to 140.0] | 108.0 [76.9 to 151.8]
  B/Brisbane (Day 21) | 785.3 [634.0 to 972.7] | 524.0 [404.9 to 678.2]

2. Primary Outcome: Number of Subjects With HI Antibody Titer Above the Cut-off Value
Description: The cut-off value assessed was ≥ 1:10 and was presented for all three vaccine influenza virus strains
Time Frame: At Day 0 and 21
Measure: Number; unit: subjects
Arm/Group | Fluarix Adult Group | Fluarix Elderly Group
Number analyzed (Participants) | 61 | 59
subjects
  A/Brisbane (Day 0) | 36 | 35
  A/Brisbane (Day 21) | 61 | 58
  A/Uruguay (Day 0) | 19 | 23
  A/Uruguay (Day 21) | 57 | 58
  B/Brisbane (Day 0) | 60 | 58
  B/Brisbane (Day 21) | 61 | 59

3. Primary Outcome: Number of Seroprotected Subjects
Description: A seroprotected subject is a subject with a serum HI antibody titer ≥ 1:40
Time Frame: At Day 0 and 21
Measure: Number; unit: subjects
Arm/Group | Fluarix Adult Group | Fluarix Elderly Group
Number analyzed (Participants) | 61 | 59
subjects
  A/Brisbane (Day 0) | 15 | 9
  A/Brisbane (Day 21) | 55 | 40
  A/Uruguay (Day 0) | 5 | 8
  A/Uruguay (Day 21) | 47 | 43
  B/Brisbane (Day 0) | 48 | 50
  B/Brisbane (Day 21) | 61 | 59

4. Primary Outcome: Number of Serconverted Subjects
Description: A seroconverted subject is a subject with a pre-vaccination serum HI titer < 1:10 and a post-vaccination serum HI titer ≥ 1:40, or a pre-vaccination serum HI titer ≥ 1:10 and a fold increase (Day 21/Day 0) ≥ 4
Time Frame: At Day 21
Measure: Number; unit: subjects
Arm/Group | Fluarix Adult Group | Fluarix Elderly Group
Number analyzed (Participants) | 61 | 59
subjects
  A/Brisbane | 44 | 30
  A/Uruguay | 44 | 39
  B/Brisbane | 39 | 30

5. Primary Outcome: Serconversion Factor
Description: Seroconversion factor, defined as the fold increase in serum HI GMT post-vaccination compared to pre-vaccination (Day 0), is presented for all three vaccine influenza virus strains
Time Frame: At Day 21
Measure: Number; unit: factor
Arm/Group | Fluarix Adult Group | Fluarix Elderly Group
Number analyzed (Participants) | 61 | 59
factor
  A/Brisbane | 12.2 | 5.9
  A/Uruguay | 12.0 | 12.4
  B/Brisbane | 7.7 | 4.9

6. Primary Outcome: Seroprotection Power
Description: Seroprotection power is defined as the number of subject who had a pre-vaccination titer < 1:40 and a post-vaccination titer ≥ 1:40
Time Frame: At Day 21
Population: Analysis was performed on the According-To-Protocol (ATP) cohort for analysis of immunogenicity, on subjects unprotected at pre-vaccination and with available results
Measure: Number; unit: subjects
Arm/Group | Fluarix Adult Group | Fluarix Elderly Group
Number analyzed (Participants) | 56 | 51
subjects
  A/Brisbane (N=46; 50) | 40 | 32
  A/Uruguay (N=56; 51) | 42 | 35
  B/Brisbane (N=13; 9) | 13 | 9

7. Secondary Outcome: Number of Subjects Reporting Solicited Symptoms
Description: Solicited local symptoms assessed include ecchymosis, induration, pain, redness, and swelling.
  Solicited general symptoms assessed include arthralgia, fatigue, headache, myalgia, shivering, sweating, and fever
Time Frame: During the 4-day (Day 0-3) post-vaccination period
Measure: Number; unit: subjects
Arm/Group | Fluarix Adult Group | Fluarix Elderly Group
Number analyzed (Participants) | 61 | 59
subjects
  Ecchymosis | 3 | 0
  Induration | 19 | 7
  Pain | 36 | 22
  Redness | 24 | 11
  Swelling | 16 | 6
  Arthralgia | 6 | 2
  Fatigue | 10 | 8
  Headache | 8 | 8
  Myalgia | 15 | 7
  Shivering | 4 | 5
  Sweating | 5 | 4
  Fever | 0 | 0

8. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AE)
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: During the 21-day (Day 0-20) post-vaccination period
Measure: Number; unit: subjects
Arm/Group | Fluarix Adult Group | Fluarix Elderly Group
Number analyzed (Participants) | 61 | 59
subjects | 7 | 6

9. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAE)
Description: An SAE is any untoward medical occurrence that: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above.
Time Frame: During the 21-day (Day 0-20) post-vaccination period
Measure: Number; unit: subjects
Arm/Group | Fluarix Adult Group | Fluarix Elderly Group
Number analyzed (Participants) | 61 | 59
subjects | 1 | 0

ADVERSE EVENTS:
Arm/Group | Fluarix Adult Group | Fluarix Elderly Group
Serious Adverse Events (participants affected / at risk) | 1/61 | 0/59
Other Adverse Events (participants affected / at risk) | 44/61 | 30/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluarix Adult Group (N=61) | Fluarix Elderly Group (N=59)
Chest pain (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fluarix Adult Group (N=61) | Fluarix Elderly Group (N=59)
Induration (General disorders) | 19 | 7
Pain (General disorders) | 36 | 22
Redness (General disorders) | 24 | 11
Swelling (General disorders) | 16 | 6
Arthralgia (General disorders) | 6 | 2
Fatigue (General disorders) | 10 | 8
Headache (General disorders) | 8 | 8
Myalgia (General disorders) | 15 | 7
Shivering (General disorders) | 4 | 5
Sweating (General disorders) | 5 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.